CLINICAL TRIAL: NCT02707406
Title: A Multi-center, Randomized, Controlled Study of Non-healing Diabetic Foot Ulcers (DFU) Treated With Standard of Care With or Without Cryopreserved Umbilical Cord Allograft (NEOX®CORD 1K)
Brief Title: Non-healing Diabetic Foot Ulcers (DFU) Treated With SoC With or Without NEOX®CORD 1K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NE-2011
Record Dates: First submitted 2016-02-25; First posted 2016-03-14 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NEOX®CORD 1K (Experimental): Intervention Other: hct/p human cell or tissue product: NEOX®CORD 1K Intervention other: human tissue application of of NEOX®CORD 1K on subject wound
  Interventions: Other: NEOX®CORD 1K; Other: standard of care
- Standard of Care (Active Comparator): Intervention Other: standard of care alone Other intervention of Standard dressing with a non-adherent wound contact layer, a classic foam pad or gauze for moderately draining wounds, a secondary bandage, and institution of an investigator-approved off-loading device
  Interventions: Other: standard of care

INTERVENTIONS:
Other: NEOX®CORD 1K — use of human tissue product wound covering
  Arms: NEOX®CORD 1K
Other: standard of care — standard wound coverings

SUMMARY:
The study is evaluating NEOX®CORD 1K, a cryopreserved human umbilical cord allograft.

The purpose of the study is to evaluate the safety, incidence and rate of wound closure following application of the product compared to standard of care in the treatment of difficult to heal diabetic foot ulcers.

DETAILED DESCRIPTION:
A total of 114 patients presenting with a non-healing diabetic foot ulcer (DFU) that is located below the malleoli (plantar only) of at least 4 weeks in duration and a size of at least 0.5 cm2 up to 5.0 cm2 for plantar wounds meeting all inclusion criteria but none of the exclusion criteria will be recruited from different trial sites. All patients will receive sharp debridement to remove non-viable tissue followed by standard of care including a sponsor approved standard dressing with a non-adherent wound contact layer, a foam pad or gauze for moderately draining wounds, a secondary bandage, and off-loading device specific to plantar wounds. Eligible patients return at two consecutive visits approximately two weeks apart to assess wound closure. Patients that exhibit a change of less than 30% reduction of the original surface area of their target wound two weeks after the screening visit following debridement will be randomized into the control group or the treatment group at this baseline visit, Week 1. The control group will continue to receive the standard of care and the treatment group will receive standard of care and NEOX® CORD 1KTM. At each weekly visit, all wounds will be adequately debrided of devitalized and necrotic tissue, and the wound dressing will be replaced. For the treatment group, application of NEOX® CORD

1KTM will be considered at each weekly treatment visit following the Investigator's assessment of wound progression. If the Investigator determines it is medically necessary, additional NEOX® CORD 1KTM will be applied, up to and including Week 12 for a maximum of no more than 10 applications. All wounds that close before Week 13 will be followed for an additional two consecutive weekly visits approximately to confirm closure before exiting the trial. Patients who experience closure at the Week 13 visit will be followed for an additional two consecutive visits up to Week 15 to confirm closure. Patients who do not experience wound closure prior to Week 13 will be considered a failure and complete the end of study/Withdrawal Visit 15 exiting the trial.

At each weekly visit, efficacy will be assessed by the extent of wound closure as determined by the wound surface area and volume measured by an electronic measurement device (Silhouette®, ARANZ Medical), after debridement if performed, using a standardized protocol. After confirmation of closure, or at Visit 15, all patients will complete the trial.

Safety will be assessed by clinical laboratory tests at screening and at End of Study/Withdrawal Visit 15, adverse event (AE) collection, and focused physical exams.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed the informed consent form
* Male or female patient at least 18 years of age or older, as of the date of the screening visit
* Confirmed diagnosis of Type I or Type II Diabetes
* Has an index ulcer that is located below the malleoli on the plantar surface of at least 0.5 cm2 or up to 5.0 cm2 when measured by the investigator staff at the screening visit using the ARANZ Silhouette post debridement.
* The depth of the index foot ulcer is graded as Wagner Grade I or II, i.e., with no evidence of exposed muscle, tendon, bone, or joint capsule
* The index ulcer is "chronic, non-healing," defined as having a duration of > 4 weeks but not > 52 weeks at the screening visit
* Arterial supply adequacy to the foot with the index ulcer confirmed by any one of the following:

Great toe pressure ≥ 40 mm/Hg

* Systolic blood pressure Ankle Brachial Index (ABI) in the range ≥ 0.65 ≤ 1.20
* TcPO2 ≥ 30 mmHg from the foot •
* Normal triphasic or biphasic waveform pattern at the ankle
* Toe Brachial Index or TBI ≥ 0.50
* Willing to follow all instructions including off-loading given by the Investigator
* Willing to return for all mandatory visits as defined in the protocol

Exclusion Criteria:

* Renal impairment marked by serum creatinine & serum total BUN > 2 times the upper limit of normal or is currently receiving renal dialysis
* Hemoglobin A1c (HbA1c) level is > 12% (108 mmol/mol)
* Has an abnormally low serum albumin, as evidenced by an albumin level ≥ 2.0 g/dl,
* A white blood cell count < 2.0 x109 /L, neutrophils < 1.0 x109 /L, platelets < 100 x109 /L
* Chronic oral steroid use of > 7.5 mg daily for greater than 7 consecutive days within the previous 30 days preceding screening
* Chronic oral or parenteral corticosteroids, or any cytotoxic agents for 7 consecutive days within the previous 30 days preceding screening,
* Has tested positive for Human Immunodeficiency Virus (HIV) or has Acquired Immune Deficiency Syndrome (AIDS)
* Has malignancy or history of cancer in 5 years preceding the screening visit other than non-melanoma skin cancer
* Pregnant women
* Women of child-bearing potential who are unwilling to avoid pregnancy or use an effective form of birth control
* Is currently enrolled or participated in another device, drug, or biological trial within 30 days of screening
* Has had within the last 7 days, is currently undergoing, or is planning for wound treatments with enzymes, growth factors, living skin, dermal substitutes including other amniotic or umbilical cord tissue therapies, or other advanced biological therapies
* Current use of topical anti-microbial or silver-containing products
* Has an allergy to primary or secondary dressing materials used in this trial
* Has an allergy to amphotericin-B or Dulbecco's Modified Eagle Medium (DMEM)
* Index ulcer is over an active Charcot deformity
* The depth of the index ulcer is graded as Wagner Grade III or higher, i.e., with evidence of exposed muscle, tendon, bone, and/or joint capsule (see Appendix 2)
* Gangrene is present on any part of the affected foot
* Current suspicion of osteomyelitis, cellulitis, or other clinical signs or symptoms of index ulcer infection
* Any previous use of NEOX® CORD 1KTM in the index ulcer

The following exclusion criteria is to be reviewed for all subjects prior to randomization:

* Has an index ulcer that has decreased in ulcer area > 30% post debridement at baseline post the Run-in period.
* Use of excluded concomitant medications, therapies, or procedures during the Run-in period.
* Clinical signs or symptoms of infection of the index ulcer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events collected throughout the trial compared between the two groups | 16 weeks

SECONDARY OUTCOMES:
Proportion of subjects in NEOX® CORD 1KTM plus standard care against standard care with complete wound closure | 12 weeks from baseline
Time in days to wound closure | 12 weeks from baseline
Proportion of subjects with complete wound closure at each of the 12 treatment | 12 weeks from baseline
Percent change in wound area (surface area cm2) at each visit compared to baseline (rate of wound closure) | up to 15 weeks from baseline
Percent change in wound volume (cm3) at each visit compared to baseline (rate of wound closure) | up to 15 Weeks from baseline
Total Number of applications of the trial product to achieve complete wound closure | up to 12 Weeks from Baseline
Difference in score of quality of life assessment determined SF-12v2 at study exit compared to baseline | up to 15 weeks from baseline
Difference in score of quality of life assessment determined by Cardiff Wound Impact Schedule (CWIS) | up to 15 weeks from baseline

CONTACTS AND LOCATIONS:
Locations (22):
- United States (19):
  - Carlsbad, California
  - Castro Valley, California
  - Fair Oaks, California
  - San Francisco, California
  - Sylmar, California
  - Washington D.C., District of Columbia
  - Miami, Florida
  - North Chicago, Illinois
  - New Orleans, Louisiana
  - Missoula, Montana
  - Las Vegas, Nevada
  - Eugene, Oregon
  - Portland, Oregon
  - Fort Worth, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Murray, Utah
  - Roanoke, Virginia
  - Virginia Beach, Virginia
- Canada (3):
  - Hamilton, Ontario
  - London, Ontario
  - Boucherville, Quebec

IPD SHARING:
Plan to Share IPD: Undecided